CLINICAL TRIAL: NCT02903875
Title: Therapeutic Education Program Aimed at Improving the Quality of Life of Laryngectomised Patients and Their Close Relatives
Brief Title: Therapeutic Education Program for Laryngectomised Patients and Their Close Relations
Acronym: PETAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: University of Lille Nord de France (Other); CERFEP CARSAT Nord-Picardie (Unknown); INSERM U1086 Cancers et Préventions (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHRC12-220
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- laryngectomised patients since 1 month: laryngectomised patients since 1 month and their close relative
  Interventions: Other: Patient therapeutic education (PTE) programme
- laryngectomised patients since 3 months: laryngectomised patients since 3 months and their close relative
  Interventions: Other: Patient therapeutic education (PTE) programme
- laryngectomised patients since 6 months: laryngectomised patients since 6 months and their close relative
  Interventions: Other: Patient therapeutic education (PTE) programme
- laryngectomised patients since 12 months: laryngectomised patients since 12 months and their close relative
  Interventions: Other: Patient therapeutic education (PTE) programme

INTERVENTIONS:
Other: Patient therapeutic education (PTE) programme

SUMMARY:
The therapeutic education of patients and their close relations is, as yet, poorly developed in France in the field of oncology, in particular for cancers of the upper aerodigestive tract. In the case of pharyngeal and laryngeal cancer, total laryngectomy associated with radiotherapy remains a reference treatment for advanced stage cancers. This mutilating surgical procedure has a major impact on the patient's life, due to its physical and functional sequelae. Its psychosocial consequences are also important, owing to the biographical disruption and the identity-related metamorphoses associated with illness and its treatment, which alter the quality of life not only of patients, but also of their close relations. Currently, care for laryngectomised patients consists essentially in informing and educating them on certain technical procedures during hospital admission. New voice education can be a long process and often involves the intervention of a speech therapist, who serves as the link between the patient and the hospital care team. These healthcare modalities often insufficiently account for the social, environmental and personal factors that interact in health-related problems.

The aim is to design, implement and evaluate a patient therapeutic education (PTE) programme, for laryngectomised patients and their close relations, aimed at improving their quality of life.

The research will be conducted over three phases:

The first phase, referred to as the "pilot" phase, will include exploratory, observational and retrospective analysis aimed at developing knowledge on the consequences of laryngectomy on the quality of life of patients and their close relations, the strengths and weaknesses of current practice in patient support and the needs expressed by the players involved (patients, relations, professional carers). This analysis will be conducted via interviews with patients and their close relations and focus groups with the healthcare professionals involved in patient care and support (hospital and independent). This first phase will enable the pluridisciplinary design of a therapeutic education programme for laryngectomised patients and their close relations which will be tested in the study's principle coordinating centre. The method defined thus is in keeping with quality criteria set by the HAS specifying that the PTE should focus on the patient, be scientifically justified, and be developed by a pluridisciplinary group reuniting representatives of patients or patient associations.

The second phase, referred to as the prospective intervention "replication" phase, aims at evaluating the programme's transferability and quality in three centres. The centres participating in this second phase already have experience in the development of PTE programmes and will be involved in the workgroup entrusted with the design of the PETAL programme during phase 1.

The third phase, referred to as the "randomised" multicentric comparative intervention phase, should enable us to assess the benefits of the developed PTE programme on the quality of life of patients and their close relations.

This is a pluridisciplinary study via which we hope to improve the quality of life of laryngectomised patients and their close relations through the design and the sustainable deployment of an innovative PTE programme in France and Belgium. This project also aims at reinforcing town-hospital links to improve help, follow-up and support for patients and their close relations, as well as dialogue between healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Patient (18-70 years) treated with total laryngectomy for cancer of the larynx, pharynx or cervical esophagus
* Patient agreeing to participate in the study (informed consent)
* Person designated as close relative by the laryngectoised patient (support person, spouse, parent, caregiver)
* Close relative agreeing to participate in the study (informed consent) after the patient himself has authorized the investigator to contact that person to offer to participate in the study
* Time since laryngectomy (group 1 : 1 month, group 2: 3 months, group 3: 6 months, group 4 : 12 months)

Exclusion Criteria:

* Physical , mental, cognitive or psychiatric disabilityof the patient to answer questions and participate in interviews and therapeutic education program
* Physical , mental, psychiatric or cognitive disability of the close relative to answer questions and participate in interviews and therapeutic education program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer of the larynx, pharynx or cervical esophagus treated with total laryngectomy and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
interview of patient and close relatives | baseline
  design, implement and evaluate a patient therapeutic education (PTE) programme, for laryngectomised patients and their close relations, aimed at improving their quality of life.

SECONDARY OUTCOMES:
transferability of patient therapeutic education (PTE) | during 1 year
  evaluating the programme's transferability in three centres
quality of patient therapeutic education (PTE) | during 1 year
  evaluating the programme's quality in three centres
quality of life (QLQC30) | baseline and 1 year after PTE
  to assess the benefits of the developed PTE programme on the quality of life of patients and their close relations

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Caen Cancer Institute, Caen
  - Caen University Hospital, Caen
  - Lille Cancer Institute, Lille
  - Lille University Hospital, Lille

IPD SHARING:
Plan to Share IPD: No